CLINICAL TRIAL: NCT02484430
Title: A Phase 2 Study of MLN0128 (TAK-228) in Relapsed and/or Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Sapanisertib in Treating Patients With Relapsed and/or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01000; NCI-2015-01000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1482; 9775 (Other: Mayo Clinic Cancer Center LAO); 9775 (Other: CTEP); N01CM00099 (NIH); UM1CA186686 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-06-29 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: B Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative; Recurrent Adult Acute Lymphoblastic Leukemia; Refractory Adult Acute Lymphoblastic Leukemia; T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sapanisertib) (Experimental): Patients receive sapanisertib PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who are non-responders and in PR at the end of course 4 may receive sapanisertib PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sapanisertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228

SUMMARY:
This phase II trial studies how well sapanisertib works in treating patients with acute lymphoblastic leukemia that has returned after a period of improvement (relapsed) or has not responded to previous treatment (refractory). Sapanisertib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete hematologic response (CR)/complete response incomplete (CRi) rate when sapanisertib (MLN0128 [TAK-228]) is administered to adult patients with relapsed/refractory acute lymphoblastic leukemia (ALL).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (CR, CRi/partial response (PR)/morphologic leukemia free state [MLFS]).

II. To determine the CR/CRi duration when MLN0128 (TAK-228) is administered to adult patients with relapsed/refractory ALL.

III. To determine the frequency of proceeding to allogeneic stem cell transplantation (SCT) for patients with relapsed/refractory ALL who achieve a response on MLN0128 (TAK-228).

IV. To determine the overall survival for relapsed/refractory ALL patients on MLN0128 (TAK-228).

TERTIARY OBJECTIVES:

I. To examine the pharmacokinetics of MLN0128 (TAK-228) in ALL patients. II. To assess whether phosphorylation of the mTOR substrate 4EBP1 decreases in leukemic blasts harvested from the bone marrow on day 8 compared to baseline.

III. To assess in an exploratory fashion whether MLN0128 (TAK-228) enhances expression of the pro-apoptotic proteins Bim and Puma in marrow ALL cells.

IV. To assess in an exploratory fashion whether Mcl-1 levels decrease in blast cells during MLN0128 (TAK-228) treatment.

V. To assess in an exploratory fashion whether a) the phospho-protein pattern at baseline or b) MLN0128 (TAK-228)-associated changes in the phospho-protein pattern differs between ALL samples that respond to therapy and those that do not.

OUTLINE:

Patients receive sapanisertib orally (PO) daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who are non-responders and in PR at the end of course 4 may receive sapanisertib PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO)-defined acute lymphoblastic leukemia and either:

  * Relapsed after achieving remission
  * Refractory to therapy
  * Newly diagnosed and ineligible for intensive chemotherapy induction Note: patients with T lineage and B lineage ALL are eligible for this trial; likewise, patients with Philadelphia chromosome positive (Ph+) (as long as they are not candidate for other therapies for Ph+) and Ph- ALL are eligible
* Bone marrow blasts of at least 10%
* At least 4 weeks away from any previous antineoplastic or investigational agent; patients may receive hydroxyurea or glucocorticoids for suppression of leukocytosis, but these must be stopped at least 24 hours (h) prior to initiation of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of > 2 months
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal
* Fasting blood glucose (FBG) < 130 mg/dL
* Hemoglobin A1C (HbA1C) < 7.0%
* Relapse after SCT is allowed but no active graft-versus-host disease (GVHD) as per treating physician; also must not exceed the number of prior induction regimens listed above; SCT does not count as line of therapy
* Negative serum pregnancy test result; Note: women of child-bearing potential and men must agree to use 1 highly effective method of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated by local labeling [e.g. United States product insert (USPI), Summary of Product Characteristics (SmPC), etc]) after the last does of study drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use highly effective barrier contraception prior to the study, for the duration of study participation, and 4 months after completion of MLN0128 (TAK-228) administration
* Ability to understand and the willingness to sign a written informed consent document
* No prior therapy with mTOR inhibitors except for rapalog treatment as part of graft-versus-host (GVH) prophylaxis or treatment
* Human immunodeficiency virus (HIV) infected patients (if HIV positive)

  * HIV infected individuals are eligible provided they meet all the protocol eligibility criteria in addition to the following:

    * No history of acquired immune deficiency syndrome (AIDS) defining illness other than a historic CD4+ T-cell nadir < 200/mm^3
    * Prior to leukemia diagnosis, the HIV disease was uncomplicated as evidenced by:

      * The CD4+ T-cell counts were generally in excess of 300/mm^3
      * The HIV viral loads were less than 200 copies/ml if on anti-HIV therapy
      * If the HIV is newly diagnosed or there is no history of using anti-HIV therapy, there are no AIDS defining conditions or other HIV-related symptoms
      * Zidovudine is not allowed as part of the anti-HIV therapy
* Patients with diabetes controlled by diet or medication are allowed on trial; controlled diabetes is defined as FBG < 130 mg/kL in the context of this study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy =< 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; treatment with glucocorticoids, hydroxyurea, and tyrosine kinase inhibitors is allowed up to 24 hour prior to initiation of therapy
* Patients with white blood cell (WBC) > 30,000 are not eligible to start therapy; however, it is permissible to use glucocorticoids and/or hydroxyurea to diminish peripheral WBC to less than 30,000 provided these agents are stopped at least 24 hours prior to the first dose of MLN0128 (TAK-228)
* Patients who are receiving any other investigational agents
* Patients with known other active cancers; skin cancers (basal or squamous) are exempted
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN0128 (TAK-228)
* There are no prohibitions of specific medications on the basis of anticipated drug-drug interactions
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; no ischemic myocardial or cerebrovascular event, placement of pacemaker, or pulmonary embolism within six months of receiving first dose of MLN0128 (TAK-228)
* Any patient receiving chronic corticosteroid administration prior to study enrollment is ineligible
* Baseline prolongation of the rate-corrected QT interval (QTc) > 480 milliseconds or history of congenital long QT syndrome or Torsades de pointes
* Concomitant administration of any proton pump inhibitor (PPI) is not permitted during the study; patients receiving PPI therapy before enrollment must stop using the PPI for 7 days before their first dose of study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aref Al-Kali, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (14):
- United States (14):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Al-Kali A, Aldoss I, Atherton PJ, Strand CA, Shah B, Webster J, Bhatnagar B, Flatten KS, Peterson KL, Schneider PA, Buhrow SA, Kong J, Reid JM, Adjei AA, Kaufmann SH. A phase 2 and pharmacological study of sapanisertib in patients with relapsed and/or refractory acute lymphoblastic leukemia. Cancer Med. 2023 Dec;12(23):21229-21239. doi: 10.1002/cam4.6701. Epub 2023 Nov 13. PMID 37960985

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Sapanisertib): Patients receive 3 mg sapanisertib PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who are non-responders and in PR at the end of course 4 may receive 3 mg sapanisertib PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Sapanisertib)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients registered were included in this analysis.
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45.5 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR or CRi)
Description: Complete response rate, defined to be a complete hematologic response (CR) or complete response incomplete (CRi) noted as the objective status at any time during treatment. A CR is defined as having less than 5% blasts in a non-hypocellular marrow with a granulocyte count of 1 x109/L (or above), and a platelet count of 100 x109/L (or higher) and absence of peripheral blood blasts with complete resolution of any extra medullary disease. A patient is defined as having a CRi if they meet all CR criteria except for residual neutropenia (ANC<1 x109/L) or thrombocytopenia (platelets<100 x109/L).
  A CR or CRi will be considered synonymous with "success". The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent exact binomial confidence intervals for the true success proportion will be calculated.
Time Frame: 61 days
Population: All patients registered and evaluated for a response were included in this analysis. One patient registered but cancelled prior to treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 15
proportion of participants | 0 [0 to 0.22]

2. Secondary Outcome: Overall Response
Description: ORR will be estimated by the total number of complete or partial responses (CR, CRi or PR), or morphologic leukemia free state [MLFS]) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
  A CR is defined as having less than 5% blasts in a non-hypocellular marrow with a granulocyte count of 1 x109/L (or above), and a platelet count of 100 x109/L (or higher) and absence of peripheral blood blasts with complete resolution of any extra medullary disease. A patient is defined as having a CRi if they meet all CR criteria except for residual neutropenia (ANC<1 x109/L) or thrombocytopenia (platelets<100 x109/L). A Partial Response (PR) is defined as the presence of trilineage hematopoiesis in the bone marrow with recovery of ANC and platelet count to above levels, but with 5-25% bone marrow blasts and ≥50% decrease in bone marrow blast percentage from baseline.
Time Frame: 61 days
Population: All patients who registered and began protocol treatment were included in this analysis. One patient registered but cancelled prior to treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 15
proportion of participants | 0 [0 to 0.22]

3. Secondary Outcome: Duration of Complete Response
Description: The distribution of duration of complete response will be estimated using the method of Kaplan-Meier.
Time Frame: 0 days
Population: Only patients who achieved a complete response were eligible for this endpoint.
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency of Proceeding to Allogeneic Stem Cell Transplantation (SCT) After Achieving Response (Complete Hematologic Response [CR]/Complete Response Incomplete [CRi] Partial Response [PR], or Morphologic Leukemia Free State [MLFS]) to Sapanisertib
Description: The frequency is estimated by the number of patients who proceed to allogeneic SCT after achieving response divided by the total number of evaluable patients who achieved a response. All evaluable patients who achieved a response will be used for this analysis. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Time Frame: 0 days
Population: Patients reporting a CR, CRi, PR or MLFS were eligible for this endpoint. No patients were analyzed because no patients achieved CR, CRi, PR or MLFS.
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: 23 months
Population: All patients registered and treated per protocol were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 15
days | 62.0 [51.0 to 155.0]

6. Secondary Outcome: Incidence of Adverse Events, Measured Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. For this endpoint, we are reporting the maximum grade adverse event per patient.
Time Frame: 91 days
Population: All participants who registered and started protocol treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sapanisertib)
Number analyzed (Participants) | 15
Participants
  Grade 3 | 0
  Grade 4 | 13
  Grade 5 | 2

ADVERSE EVENTS:
Time Frame: All cause mortality was followed for 23 months and adverse events were followed for 6 months.
Description: All patients were included in this section.
Arm/Group | Treatment (Sapanisertib)
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sapanisertib) (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sapanisertib) (N=16)
Anemia (Blood and lymphatic system disorders) | 9 (37)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anal mucositis (Gastrointestinal disorders) | 1 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (9)
Fever (General disorders) | 1 (2)
Gait disturbance (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Activated partial throm time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (4)
Creatinine increased (Investigations) | 2 (2)
Fibrinogen decreased (Investigations) | 1 (5)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (7)
Neutrophil count decreased (Investigations) | 5 (9)
Platelet count decreased (Investigations) | 7 (26)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Lethargy (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT02484430/Prot_SAP_000.pdf